CLINICAL TRIAL: NCT03070626
Title: Preoperative Loading With Carbohydrates in Lung Cancer Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Per Reidar Woldbæk, MD, PhD, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2016/2020
Record Dates: First submitted 2017-01-20; First posted 2017-03-03 (Actual); Last update posted 2017-03-27 (Actual); Status verified 2017-03

CONDITIONS: Lung Neoplasm
Keywords: General Surgery; Carbohydrates; Perioperative
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional group (Experimental): Carbohydrate-rich, dietary supplement: PreOp® 800ml day before surgery and PreOp® 400ml 2-4hours preoperative.
  Interventions: Dietary Supplement: PreOp®
- Control group (No Intervention): Standard of care: Fasting from 24hours (midnight), night before surgery.

INTERVENTIONS:
Dietary Supplement: PreOp® — No preoperative drink.
  Other Names: NutriciaPreOp®
  Arms: Interventional group

SUMMARY:
Administration of preoperative oral carbohydrates are suggested to reduce insulin resistance due to surgical stress.

The aim of this study is to investigate whether preoperative oral carbohydrate loading can contribute to lower incidence of postoperative discomfort and to reduce complications in elective lung cancer patients undergoing video assisted thorascopic surgery (VATS).

DETAILED DESCRIPTION:
Fasting from 6-12hours before elective surgery is still standard of care in many departements, including our departement in Oslo University Hospital.

Surgery is a trauma that triggers a catabolic stress response with high emissions of hormones and immune activation. These activations can affect brain, heart, muscles and liver. The metabolic changes may in addition influence development of pain, tissue damage, ileus, tachycardia and other hemodynamic disturbances. Preoperative fasting has shown an increase of surgical stress and to impact catabolic processes which secondarily may lead to insulin resistance and hyperglycemia in non-diabetic patients. Insulin resistance and hyperglycaemia are known to increase the incidence of postoperative infections. Previous studies have also shown that prolonged fasting increases the incidence of gastrointestinal problems. A 12 hour fast before surgery has shown delayed recovery.

Studies have shown that patients undergoing lung cancer surgery suffer from multiple symptoms and experience discomfort in the postoperative phase. Symptoms include dyspnea, fatigue, pain, weakness, cough, dry mouth, nervousness, difficulty sleeping, stomach-/intestinal-problems and lack of appetite. Carbohydrate-rich supplements have shown a positive effect on other perioperative symptoms and measures, but is to our knowledge currently not investigated in lung cancer surgery.

Therefore, there is a need to explore the possible advantages of preoperative oral carbohydrate loading in lung cancer surgery.

The primary aim of this study is to investigate whether preoperative carbohydrate loading with PreOp® provides less postoperative discomfort in the early postoperative phase measured by Quality of Recovery-40 (QoR-40), a validated and widely used measure of quality of recovery.

The secondary aim is to investigate if preoperative loading with carbohydrates affect the incidence of postoperative complications such as stomach-/intestinal problems and heart rhythm disorder, in addition to contribute to faster mobilization and to reduce hospital length of stay.

This study may provide important data regarding the lung cancer patients perioperative symptoms, complications and well-being when using a carbohydrate-rich supplement as intervention to standard of care.

In this study, the intervention group will be given 800ml of a oral carbohydrate supplement, PreOp®, the night before surgery and 400ml of the same supplement, PreOp®, 2-4 hours prior to surgery. The control group will be fasted from 24h, the night before surgery, in accordance to the departements standard of care.

Both groups, the interventional and the control group, will follow the department's perioperative course with regard to anesthetic and surgical procedures.

ELIGIBILITY:
Inclusion Criteria:

adult patients undergoing elective video-assisted thoracoscopic surgery due to lung neoplasms.

* ability to understand and speak Norwegian

Exclusion Criteria:

* impaired gastric emptying
* diabetes
* ongoing treatment for pain
* ongoing infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2017-03-20 (Actual); Primary Completion 2020-01 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative discomfort measured by the questionnaire "Quality of recovery 40" (QoR-40) measured on the first postoperative day. | First postoperative day
  Postoperative discomfort measured by the questionnaire "Quality of recovery 40" (QoR-40) measured on the first postoperative day.

SECONDARY OUTCOMES:
Gastrointestinal discomfort postoperatively. | First seven postoperative days.
  Number of patients experiencing nausea, vomiting, diarrhea and/or obstipation.
Heart rhythm disturbances postoperatively. | First seven postoperative days.
  Number of patients with arrhythmia lasting more than 5 min or treated with antiarrhythmic agents.
Time to mobilization. | First seven postoperative days.
  Time to mobilization out of bed (to chair or walking) as registered by the attending nurse.
Length of stay | First seven postoperative days.
  Length of hospital stay to discharge for index admission.

CONTACTS AND LOCATIONS:
Locations (1):
- Oslo University Hospital, Oslo, Oslo County, Norway

IPD SHARING:
Plan to Share IPD: No